CLINICAL TRIAL: NCT01233063
Title: Diet and Activity Promotion Among Older Working Adults
Acronym: ALIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Berkeley Analytics, Inc. (Industry)
Responsible Party: Principal Investigator, Gladys Block, Scientific Director, Berkeley Analytics, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5R44AG032241-03 (NIH)
Record Dates: First submitted 2010-10-27; First posted 2010-11-03 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Cardiovascular Disease; Diabetes; Obesity; Aging
Keywords: behavior change; physical activity; nutrition; fruits and vegetables; saturated fat; trans fat; added sugars; email; web; obesity; aging
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alive2 (Experimental): Lifestyle Intervention delivered via email and web
  Interventions: Behavioral: Physical Activity and Diet Intervention via Alive2
- Alive2 plus automated phone/print (Experimental): All of Arm 1 components, plus biweekly tailored automated phone coaching plus monthly tailored automated print materials.
  Interventions: Behavioral: Physical Activity and Diet Intervention via Alive2
- Control (Placebo Comparator): Monthly emailed newsletter on other aspects of wellness, excluding diet and physical activity
  Interventions: Behavioral: Physical Activity and Diet Intervention via Alive2

INTERVENTIONS:
Behavioral: Physical Activity and Diet Intervention via Alive2 — Weekly email/web goal-setting intervention to improve physical activity and diet, with and without additional phone and mail support.

SUMMARY:
The trial will test whether the Alive email-delivered health behavior program can improve subjects' physical activity, fruits and vegetables and saturated/trans fats and added sugars.

ELIGIBILITY:
Inclusion Criteria:

* aged 50+
* currently employed
* access to email/web

Exclusion Criteria:

* angina

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in physical activity | 3, 6, 9, 12 months
  Change in physical activity as reported on questionnaire
Change in Fruits and Vegetables | 3, 6, 9, 12 months
  Change in fruits and vegetables as reported on questionnaire
Change in saturated fats | 3, 6, 9, 12 months
  Change in saturated fat intake as reported on questionnaire
Change in added sugar | 3, 6, 9, 12 months
  Change in added sugar as reported on questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gladys Block, PhD, Principal Investigator — Berkeley Analytics, Inc.
Locations (1):
- Berkeley Analytics, Inc., Berkeley, California, United States